CLINICAL TRIAL: NCT04827121
Title: Transmuscular Quadratus Lumborum Block Versus Supra-inguinal Fascial Iliac Compartment Block for Total Hip Arthroplasty: a Randomized, Prospective Study
Brief Title: Comparison of Fascial Iliac Compartment Block and Quadratus Lumborum Block for Hip Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wei Mei, Deputy Director of Anesthesiology Department of Tongji Hospital Affiliated to Huazhong University of Science and Technology, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TJ-IRB20210141
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Analgesia
Keywords: Ultrasound; Total hip arthroplasty; Nerve block
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fascial iliac compartment block group (Active Comparator): Patients in this group will recieve supra-inguinal fascial iliac compartment block after anesthesia induction.
  Interventions: Procedure: Fascial iliac compartment block
- Quadratus lumborum block group (Active Comparator): Patients in this group will recieve quadratus lumborum block after anesthesia induction.
  Interventions: Procedure: Quadratus lumborum block

INTERVENTIONS:
Procedure: Fascial iliac compartment block — Patients will recieve supra-inguinal approach of fascial iliac compartment block under ultrasound guidance with 30 ml of 0.5 percent ropivacaine.
  Arms: Fascial iliac compartment block group
Procedure: Quadratus lumborum block — Patients will recieve transmuscular approach of quadratus lumborum block under ultrasound guidance with 30 ml of 0.5 percent ropivacaine.
  Arms: Quadratus lumborum block group

SUMMARY:
Iliac fascia block has a long history of analgesia in patients with hip fractures. A large number of clinical studies have confirmed its efficacy, and there are also randomized controlled studies supporting its effectiveness in analgesia after total hip replacement surgery.Quadratus lumborum block is a new block technique developed in last decade, and there are also a few randomized controlled studies supporting its effectiveness in postoperative analgesia for total hip replacement.The purpose of the present study was to find out whether these two different approaches of fascial compartment block have similar effects on postoperative analgesia after total hip replacement.

ELIGIBILITY:
Inclusion Criteria:

* ASA class 1-3
* BMI between 20-36kg/m^2
* Scheduled to undergo total hip replacement

Exclusion Criteria:

* A history of chronic opioids or steroid consumption
* Coagulapathy or anticoagulation
* Pregnancy
* Allergic to local anesthetics Neurological dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative opioids consumption at 24 hours | Within 24 hours
  Cumulative consumption of sufentanil from PCA device at 24 hours after surgery

SECONDARY OUTCOMES:
NRS score with movement at 6,12,and 24 hours | at 6,12,and 24 hours
  Patients' NRS score with movement at 6,12,and 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Wei Mei, PhD, Principal Investigator — Tongji Hospital
Locations (1):
- Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No